CLINICAL TRIAL: NCT03863028
Title: Development and Validation of a Simulator-based Test in Transurethral Resection of Bladder Tumors
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Sarah Hjartbro Bube, MD, Ph.D. student, Zealand University Hospital
Other Study IDs: 17-000048
Record Dates: First submitted 2019-03-01; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Validity-evidence for a Simulator-based Test; Virtual Simulation; Bladder Cancer; Surgical Skill Training; Medical Education; Transurethral Resection of Bladdertumors
Keywords: Validity-evidence; TURB; Mastery Learning; Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Novice: Residents with no individual experience in TUR-B defined as no prior hands-on surgical experience in TURB
  Interventions: Other: Simulation training
- Intermediates: Residents who have performed 10 to 30 TURBs.
  Interventions: Other: Simulation training
- Experienced: Consultants with experience in the procedure defined as more than 100 TURBs.
  Interventions: Other: Simulation training

INTERVENTIONS:
Other: Simulation training — It is not a randomized trial - all three groups are exposed to simulation training.

SUMMARY:
Bladder cancer (BC) is the seventh most common cancer in men worldwide and fourth most common cancer among Danish men. BC is estimated to be the most cost expensive cancer pr. patient life. BC is diagnosed, staged and if possible treated with a transurethral bladder tumor resection (TUR-B).

The prognosis of BC is depending on the depth of invasion, which makes the quality of the TURB procedure of utmost importance. Retrospective studies from Sweden and Canada on resident involvement in TURB procedures indicated that the TURBs were insufficient with regard to staging and had a higher need of repeating TURB.

Surgical training for TURB in Denmark today is based on the Halstedian principle: "See one, do one, teach one", comparable to training in Sweden and Canada. Thus, there is a need to develop better and safer principles for training.

Simulators for surgical procedures have a promising role in the surgical training. The project will explore the effect of simulation training on the quality in transurethral resection of bladder tumors.

Based on our findings the principles of simulator training will be integrated in a curriculum for simulator-based TURB training for urological surgeons in Denmark.

The collaboration research group is composed of medical doctors in urological surgery at Urological Department at Zealand University Hospital, Roskilde (ROS) and experts in medical simulation at Copenhagen Academy for Medical Education and Simulation at Rigshospitalet (CAMES).

DETAILED DESCRIPTION:
The incidence of bladder tumors is increasing and is more than 2,000 in Denmark. The bladder tumor is initially treated by transurethral resection (TURB) classifying the tumor by debt of invasion. The bladder wall is composed of urothelium, lamina propria and muscularis propria also known as the detrusor muscle. Bladder cancer (BC), defined as detrusor-muscle invasive tumors, are found in approximately 50% of bladder tumors. BC is the seventh most common cancer disease among men worldwide, and the fourth most common cancer in men in Denmark. Superficial bladder tumors can be treated with TURB whereas BC is treated with radical cystectomy. Thus, it is of utmost importance that TURB is done with sufficient resection of the detrusor muscle to ensure that the patient is staged correctly to optimise treatment.

TURB was first described and performed by Desormeaux in 1867 and the obstacles for the surgeon remain the same more the 150 years after. TUR-B demands haptic skills, the ability to identify the layers of the bladder wall, the ability to perceive the stiffness of the tissue through radial and tangential movements and the ability to translate two-dimensional pictures to a three-dimensional understanding and at the same time move surgical instruments around an axis.

As TUR-B is performed through the urethra with one scope only, the learner is left with observation of the master until the day occurs where the learner is trusted the scope. Thus, the gap between seeing and doing TURB remains significant.

The outcome of TURB have been shown to be dependent on surgeon-experience, with a higher risk for insufficient resections with lower surgeon experience. A recent Canadian study from a single centre showed that resident involvement in TUR-B had fewer complete resections including the detrusor muscle layer in the pathological specimen and patients had delayed time to cystectomy when compared to patients who had the TUR-B performed by attending urologists. Thus, both patient safety and quality of care are compromised when residents are involved in the treatment and staging of patients with bladder tumors.

The current education in TURB in Denmark is based on classical apprenticeship as it has been for the last 150 years, with the resident learning from a supervisor while performing TURB on patients.

Needs assessment analyses among specialists in urology and medical education in Denmark in 2017 identified TURB as a procedure in which simulation based skill acquisition are desired.

Simulation-based training is increasingly used in medical education. The opportunity to train a procedure repeatedly in a secure, stress-free environment with several different scenarios is appealing. Even though simulation-based training carries these promising opportunities, the challenge, when introducing simulation-based training, is to identify if the training transfer to actually improved performance on patients. Thus, we need to test if the simulator training leads to a level of minimum competency before progressing to performance on patients. A minimum passing standard should not be defined by amount of training, but by simulator performance outcomes.

Thus, we need to define test outcomes that identify competency before introducing a simulation-based test. Mastery learning (ML) is an educational theory in which the learner is to train until reaching a minimum acquisition level. The endpoint of the training is hereby a predefined competency level, and not an arbitrary amount of training hours. In the light of the ML framework the principle of directed self-regulated learning (DSRL) has evoked. DSRL is a learning-approach where the student regulates his/her own progress through a defined training protocol without guidance from an instructor. The theory is that this approach provides the student the opportunity to develop own strategies and to learn from mistakes, while also increasing the availability of training independent of supervision from a busy faculty.(20) DSRL can be modified to ensure that the learner do not learn unappropriated methods by either written theoretical material, video instructions, a non-expert assistant or all of them. Thus, the purpose of this trial is to develop and gather validity evidence for a simulator-based test in TURB based on the principles of ML and DSRL.

Hypothesis Overall: A simulator-based test can identify competency-levels with regard to a score based simulator metrics.

Aim of project To develop and gather validity evidence for a simulator-based test in TURB.

Research Question

* Can the test discriminate between varying competency levels?
* Can we establish a level of competency by a test in simulator-based TURB training?

ELIGIBILITY:
Inclusion Criteria:

* Novice: Residents with no individual experience in TUR-B defined as no prior hands-on surgical experience in TURB.
* Intermediates: Residents who have performed 10 to 30 TURBs.
* Experienced: Consultants with experience in the procedure defined as more than 100 TURBs.
* All participants: Reasonable Danish skills and must give informed written consent to participate.

Exclusion Criteria:

* Exclusion criteria for all participants: Prior systematic experience on the Simbionix/VirtaMed UroSimTM simulator.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Based on previous studies on TURB simulation and surgeon depending surgical outcomes, three groups are conducted: Residents with no individual experience in TUR-B defined as no prior hands-on surgical experience in TURB, intermediary experienced senior residents defined as surgeons who have performed between 10 and 30 TURBs and consultants with expertise in the procedure defined as more than 100 TURBs.(6,16,21,22) Residents, intermediates, and consultants at the three Urological Departments of the Zealand Region and the Capital Region will be invited to voluntary participation by written invitation. All eligible doctors will be categorised in the three groups until the sample size is reached.
Sampling Method: Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Mean test score | Through study completion, an average of 4 weeks
  Based on simulator metrics with significant discriminatory ability between different experience levels, a test score is constructed.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Copenhagen Academy for Medical Education and Simulation, Copenhagen, Danmark
  - Urology Department, Zealand University Hospital, Roskilde

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allard CB, Meyer CP, Gandaglia G, Chang SL, Chun FK, Gelpi-Hammerschmidt F, Hanske J, Kibel AS, Preston MA, Trinh QD. The Effect of Resident Involvement on Perioperative Outcomes in Transurethral Urologic Surgeries. J Surg Educ. 2015 Sep-Oct;72(5):1018-25. doi: 10.1016/j.jsurg.2015.04.012. Epub 2015 May 21. PMID 26003818
- [Background] Bos D, Allard CB, Dason S, Ruzhynsky V, Kapoor A, Shayegan B. Impact of resident involvement in endoscopic bladder cancer surgery on pathological outcomes. Scand J Urol. 2016 Jun;50(3):234-8. doi: 10.3109/21681805.2016.1163616. Epub 2016 Apr 4. PMID 27045233
- [Background] Amin MB, Smith SC, Reuter VE, Epstein JI, Grignon DJ, Hansel DE, Lin O, McKenney JK, Montironi R, Paner GP, Al-Ahmadie HA, Algaba F, Ali S, Alvarado-Cabrero I, Bubendorf L, Cheng L, Cheville JC, Kristiansen G, Cote RJ, Delahunt B, Eble JN, Genega EM, Gulmann C, Hartmann A, Langner C, Lopez-Beltran A, Magi-Galluzzi C, Merce J, Netto GJ, Oliva E, Rao P, Ro JY, Srigley JR, Tickoo SK, Tsuzuki T, Umar SA, Van der Kwast T, Young RH, Soloway MS. Update for the practicing pathologist: The International Consultation On Urologic Disease-European association of urology consultation on bladder cancer. Mod Pathol. 2015 May;28(5):612-30. doi: 10.1038/modpathol.2014.158. Epub 2014 Nov 21. PMID 25412849
- [Background] Ploeg M, Aben KK, Kiemeney LA. The present and future burden of urinary bladder cancer in the world. World J Urol. 2009 Jun;27(3):289-93. doi: 10.1007/s00345-009-0383-3. Epub 2009 Feb 15. PMID 19219610
- [Background] Jancke G, Rosell J, Jahnson S. Impact of surgical experience on recurrence and progression after transurethral resection of bladder tumour in non-muscle-invasive bladder cancer. Scand J Urol. 2014 Jun;48(3):276-83. doi: 10.3109/21681805.2013.864327. Epub 2013 Nov 29. PMID 24286506
- [Background] Mariappan P, Zachou A, Grigor KM; Edinburgh Uro-Oncology Group. Detrusor muscle in the first, apparently complete transurethral resection of bladder tumour specimen is a surrogate marker of resection quality, predicts risk of early recurrence, and is dependent on operator experience. Eur Urol. 2010 May;57(5):843-9. doi: 10.1016/j.eururo.2009.05.047. Epub 2009 Jun 6. PMID 19524354
- [Background] Nisky I, Huang F, Milstein A, Pugh CM, Mussa-Ivaldi FA, Karniel A. Perception of stiffness in laparoscopy - the fulcrum effect. Stud Health Technol Inform. 2012;173:313-9. PMID 22357009
- [Background] Gallagher AG, McClure N, McGuigan J, Ritchie K, Sheehy NP. An ergonomic analysis of the fulcrum effect in the acquisition of endoscopic skills. Endoscopy. 1998 Sep;30(7):617-20. doi: 10.1055/s-2007-1001366. PMID 9826140
- [Background] Mariappan P, Finney SM, Head E, Somani BK, Zachou A, Smith G, Mishriki SF, N'Dow J, Grigor KM; Edinburgh Urological Cancer Group. Good quality white-light transurethral resection of bladder tumours (GQ-WLTURBT) with experienced surgeons performing complete resections and obtaining detrusor muscle reduces early recurrence in new non-muscle-invasive bladder cancer: validation across time and place and recommendation for benchmarking. BJU Int. 2012 Jun;109(11):1666-73. doi: 10.1111/j.1464-410X.2011.10571.x. Epub 2011 Nov 1. PMID 22044434
- [Background] Herr HW, Donat SM. Quality control in transurethral resection of bladder tumours. BJU Int. 2008 Nov;102(9 Pt B):1242-6. doi: 10.1111/j.1464-410X.2008.07966.x. No abstract available. PMID 19035888
- [Background] Richterstetter M, Wullich B, Amann K, Haeberle L, Engehausen DG, Goebell PJ, Krause FS. The value of extended transurethral resection of bladder tumour (TURBT) in the treatment of bladder cancer. BJU Int. 2012 Jul;110(2 Pt 2):E76-9. doi: 10.1111/j.1464-410X.2011.10904.x. Epub 2012 Feb 7. PMID 22313727
- [Background] Miladi M, Peyromaure M, Zerbib M, Saighi D, Debre B. The value of a second transurethral resection in evaluating patients with bladder tumours. Eur Urol. 2003 Mar;43(3):241-5. doi: 10.1016/s0302-2838(03)00040-x. PMID 12600426
- [Background] Naselli A, Hurle R, Paparella S, Buffi NM, Lughezzani G, Lista G, Casale P, Saita A, Lazzeri M, Guazzoni G. Role of Restaging Transurethral Resection for T1 Non-muscle invasive Bladder Cancer: A Systematic Review and Meta-analysis. Eur Urol Focus. 2018 Jul;4(4):558-567. doi: 10.1016/j.euf.2016.12.011. Epub 2017 Jan 13. PMID 28753839
- [Background] Nayahangan LJ, Bolling Hansen R, Gilboe Lindorff-Larsen K, Paltved C, Nielsen BU, Konge L. Identifying content for simulation-based curricula in urology: a national needs assessment. Scand J Urol. 2017 Dec;51(6):484-490. doi: 10.1080/21681805.2017.1352618. Epub 2017 Jul 26. PMID 28743217
- [Background] Aydin A, Ahmed K, Shafi AM, Khan MS, Dasgupta P. The role of simulation in urological training - A quantitative study of practice and opinions. Surgeon. 2016 Dec;14(6):301-307. doi: 10.1016/j.surge.2015.06.003. Epub 2015 Jul 4. PMID 26148761
- [Background] Aydin A, Raison N, Khan MS, Dasgupta P, Ahmed K. Simulation-based training and assessment in urological surgery. Nat Rev Urol. 2016 Sep;13(9):503-19. doi: 10.1038/nrurol.2016.147. Epub 2016 Aug 23. PMID 27549358
- [Background] Brydges R, Nair P, Ma I, Shanks D, Hatala R. Directed self-regulated learning versus instructor-regulated learning in simulation training. Med Educ. 2012 Jul;46(7):648-56. doi: 10.1111/j.1365-2923.2012.04268.x. PMID 22691145